CLINICAL TRIAL: NCT05469880
Title: Evaluation of the Efficacy and Tolerance of Formula 609613 37 in Acneic Patients as an Adjunct to and in Addition to 5% Benzoyl Peroxide for 6 Months
Brief Title: Efficacy and Tolerance of Formula 609613 37 in Acneic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRP09001-EFFACLAR DUO
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Acne
Keywords: acne; lipohydroxyacid; salicylic acid; benzoyl peroxide; dermocosmetic
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The creams are packaged in white tubes with specific labelling that does not allow to identify them. The 5% benzoyl peroxide tubes are delivered in commercial form.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moisturizing cream and 5% benzoyl peroxide gel (Active Comparator): Participants apply the 5% benzoyl peroxide gel every evening and the moisturizing cream every morning for 3 months. Then they are divided into 2 groups: one applies the anti-acne face cream every morning for 3 months and the other one the moisturizing cream every morning for 3 months.
  Interventions: Other: moisturizing cream and 5% benzoyl peroxide gel
- anti-acne face cream and 5% benzoyl peroxide gel (Experimental): Participants apply the 5% benzoyl peroxide gel every other night and the anti-acne face cream every morning for 3 months. Then they are divided into 2 groups: one applies the anti-acne face cream every morning for 3 months and the other one the moisturizing cream every morning for 3 months.
  Interventions: Other: anti-acne face cream and 5% benzoyl peroxide gel

INTERVENTIONS:
Other: moisturizing cream and 5% benzoyl peroxide gel — Group A: Eclaran 5% every evening and formula 609567 49 every morning, for 3 months.
  Then the group is divided: Group A1/ formula 609613 37 and Group A2/ formula 609567 49 every morning, for the next 3 months
  Arms: moisturizing cream and 5% benzoyl peroxide gel
Other: anti-acne face cream and 5% benzoyl peroxide gel — Group B: Eclaran 5% every other night and 609613 37 every morning, for 3 months.
  Then the group is divided: Group B1/ 609613 37 and Group B2/ formula 609567 49 every morning, for the next 3 months
  Arms: anti-acne face cream and 5% benzoyl peroxide gel

SUMMARY:
Acne affects most adolescents and young adults with varying severity and presentation. For early or localized forms, the first-line treatment is usually local. The available treatments often lead to local irritation, particularly during the first few weeks of use. This is why creams containing exfoliating agents have long been used in acne, as they are considered to allow a faster disappearance of superficial lesions.

The objective of this 6-month double-blind study is to demonstrate in 100 acneic patients the interest of an anti-acne face cream as an adjunct to and in addition to a 5% benzoyl peroxide gel.

DETAILED DESCRIPTION:
The study is conducted in accordance with the protocol and the legislative and regulatory provisions in force (after obtaining authorization of the French health authorities and the favorable opinion of the ethics committee).

Regarding the statistical analysis, two different analysis are performed:

* Descriptive analysis: quantitative variables are described by the mean and standard deviation and qualitative variables by the raw number of each modality and the corresponding percentage.
* Comparative analysis: for quantitative variables, inter-group comparisons are made by a Student's T-test or a non parametric Mann-Whitney test if necessary. For qualitative variables, comparisons are made using a Chi-square test, if the expected number of participants is less than 5, Fischer's exact test on a 4-box contingency tables is used.

A significant level of p <0.05 is considered as significant. A double-data entry is carried out then a comparison of the two databases is performed. Finally internal and external consistency tests are planned. Missing data are described and possibly analyzed.

ELIGIBILITY:
Inclusion Criteria:

* acneic facial skin
* between 20 and 50 non-inflammatory lesions on the face
* between 10 and 40 superficial inflammatory lesions on the face
* no local acneic treatment in the previous 15 days
* no treatment with isotretinoin in the previous 3 months
* agreeing to apply only the study products

Exclusion Criteria:

* less than 20 or more than 50 non-inflammatory lesions on the face
* less than 10 or more than 40 superficial inflammatory lesions on the face
* prescription of a local acne treatment for less than 15 days
* prescription of an antibiotic treatment for less than 1 month
* prescription of an isotretinoin treatment for less than 3 months
* changing toiletries and hygiene products regularly

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10-21 (Actual); Primary Completion 2010-05-25 (Actual); Study Completion 2010-05-25 (Actual)

PRIMARY OUTCOMES:
change in the composite score | from baseline to month 6
  the investigator evaluates i) the skin sensitivity (erythema, desquamation) and ii) the global tolerance on a 4-point scale (i) from Absent to Important and ii) from Nil to Excellent)

SECONDARY OUTCOMES:
change in the lesion count | from baseline to month 6
  counting of non-inflammatory (open and closed comedones) and inflammatory (papules, pustules) lesions
change in the evaluation of skin sensitivity by the patient | from baseline to month 6
  evaluation of the skin sensitivity (pruritus, tingling sensation, burning sensation) on a 4-point scale (from Absent to Important)
change in the evaluation of global tolerance by the patient | from baseline to month 6
  evaluation on a 4-point scale (from Nil to Excellent)
change in the evaluation of the efficacy by the investigator and patient | from baseline to month 6
  evaluation on a 4-point scale (from Nil to Excellent)
change in the evaluation of the global efficacy by the investigator | from baseline to month 6
  evaluation on a 6-point scale (from No lesion to Very severe)
change in the quality of life | from baseline to month 6
  evaluation of the quality of life of patients with the Cardiff Acne Disability Index (CADI) score